CLINICAL TRIAL: NCT07276763
Title: Impact of Discontinuing GLP-1 Receptor Agonists for Two Weeks Prior to Upper Endoscopy on the Risk of Gastric Retention: A Retrospective Observational Study
Brief Title: Impact of Discontinuing GLP-1 Receptor Agonists for Two Weeks Prior to Upper Endoscopy on the Risk of Gastric Retention
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2025K368
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Gastric Retention
Keywords: Glucagon-like peptide-1 receptor agonists; Gastric Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No GLP-1RA group: Patients with no prescription record of GLP-1RAs, or whose most recent prescription was more than 3 months before the EGD
  Interventions: Other: No Intervention: Observational Cohort
- GLP-1RA Continued group: Patients who met both of the following criteria:
  1. Continued use of a GLP-1RA (e.g., semaglutide or dulaglutide) within 3 months prior to EGD;
  2. Underwent painless EGD before August 2024, when our institution had not yet implemented restrictions on GLP-1RA use for painless endoscopy.
  Interventions: Other: No Intervention: Observational Cohort
- GLP-1RA Held 2 Weeks group: Patients who met both of the following criteria:
  1. Continued use of a GLP-1RA (e.g., semaglutide or dulaglutide) within 3 months prior to EGD;
  2. Underwent painless EGD after August 2024, when institutional policy mandated that patients discontinue GLP-1RAs for at least 14 days prior to painless EGD.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
A retrospective observational study to explore the impact of discontinuing GLP-1 receptor agonists for two weeks prior to upper endoscopy on the risk of gastric retention

DETAILED DESCRIPTION:
Glucagon-like peptide-1 receptor agonists (GLP-1RAs), including semaglutide, liraglutide, and dulaglutide, are widely used for the management of type 2 diabetes and obesity. These agents improve glycemic control in part by delaying gastric emptying, but this pharmacologic effect may increase the risk of retained gastric contents (RGC) and aspiration during anesthesia or sedation. In 2023, the American Society of Anesthesiologists (ASA) and the American Society for Gastrointestinal Endoscopy (ASGE) issued recommendations to withhold GLP-1RAs before procedures; however, the optimal discontinuation interval remains uncertain.

Using the electronic medical record system of Huadong Hospital, this retrospective study analyzed patients who underwent upper endoscopy between August 2023 and May 2025 to examine the association between different GLP-1RA exposure patterns and the risk of RGC, providing evidence to inform optimization of pre-procedural discontinuation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective upper endoscopy
* Complete clinical information available, including endoscopy report, age, sex, BMI, history of diabetes, prior gastric surgery, and gastrointestinal symptom

Exclusion Criteria:

* Presence of upper gastrointestinal malignancy or obstruction
* History of gastric surgery (including ESD, gastrectomy, gastric bypass, etc.)
* Emergency endoscopy or non-elective procedures
* Missing key clinical information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent elective EGD at Huadong Hospital and had complete retrievable information on medication use, medical records, and endoscopy reports
Sampling Method: Non-Probability Sample
Enrollment: 16509 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of gastric retention | Immediately at study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)